CLINICAL TRIAL: NCT00035282
Title: A Double-Blind, Placebo- and Active-Controlled Acute and Extension Study of MK0869 in the Treatment of Patients With Major Depressive Disorder
Brief Title: Treatment of Patients With Major Depressive Disorder With MK0869 (0869-060)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0869-060; Formally-103; 2006_401
Record Dates: First submitted 2002-05-02; First posted 2002-05-03 (Estimated); Last update posted 2015-02-09 (Estimated); Status verified 2015-02

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Aprepitant

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: aprepitant
  Other Names: MK0869
Drug: Comparator: placebo (unspecified)

SUMMARY:
A clinical study to determine the efficacy and safety of an investigational medication (MK0869) in the treatment of depression.

DETAILED DESCRIPTION:
The duration of treatment is 8 weeks.

ELIGIBILITY:
Patients with Major Depressive Disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2001-09; Primary Completion 2003-12 (Actual); Study Completion 2003-12 (Actual)

PRIMARY OUTCOMES:
HAMD-17 total score at week 8. Tolerability. | at week 8

SECONDARY OUTCOMES:
CGI-I score at week 8, at least 50% reduction in the HAMD-17 total score, and Sheehan Disability Score at Week 8 | at week 8

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Liu KS, Snavely DB, Ball WA, Lines CR, Reines SA, Potter WZ. Is bigger better for depression trials? J Psychiatr Res. 2008 Jul;42(8):622-30. doi: 10.1016/j.jpsychires.2007.07.003. Epub 2007 Sep 7. PMID 17825841